CLINICAL TRIAL: NCT03588754
Title: Does Propranolol, a Beta Blocker, Attenuate Stress-Induced Drinking?
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000022090; R01AA022285 (NIH); 1U54AA027989-01 (NIH)
Record Dates: First submitted 2018-07-03; First posted 2018-07-17 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol (Experimental): Propranolol extended release (160mg/day). Administered orally once daily at 10:00PM. Titration schedule Days 1-3 60mg, Days 4-7 80mg, Days 8-11 120mg, and Days 12-14 160mg until steady state.
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Administered orally once daily at 10:00PM
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Propranolol Extended Release (160mg/day).
  Arms: Propranolol
Drug: Placebo — Placebo pill administered orally.
  Arms: Placebo

SUMMARY:
For this protocol, the investigators plan to conduct a pilot study evaluating the effect of propranolol on alcohol consumption. Using a parallel design, the investigators plan to randomize 20 non-treatment seeking adults with alcohol use disorders (DSM-5) to propranolol extended release (160mg/day or placebo; n=10 per cell) to evaluate whether propranolol reduces alcohol self-administered in the laboratory. Importantly, the investigators will evaluate whether propranolol counteracts stress-induced effects on alcohol self-administration. Following titration to steady state medication levels over a 2-week period, each subject will complete two laboratory sessions consisting of a well validated method for inducing stress or neutral/relaxing state (order counterbalanced), followed by a 2-hour alcohol self-administration paradigm known to be sensitive to medication effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65
2. Able to read and write English
3. Meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for current (past 6 months) alcohol use disorders
4. Able to take oral medications and willing to adhere to medication regimen

Exclusion Criteria:

1. Participants with any significant current medical conditions.
2. Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD)
3. Suicidal, homicidal or evidence of current (past 6-month) mental illness.
4. Specific exclusions for administration of propranolol not already specified.
5. Subjects likely to exhibit clinically significant alcohol withdrawal during the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption | 120 minutes
  Mean mls of alcohol consumed (maximum of 120 mg/dL) for propranolol and placebo groups during 120 minute alcohol self administration sessions taking place as close to Day 15 and Day 19 as possible of medication dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry McKee, PhD, Principal Investigator — Professor
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No